CLINICAL TRIAL: NCT04563065
Title: Active Pregnancy, Prevention Against the Effects of COVID-19
Brief Title: Active Pregnancy Against COVID-19
Acronym: ACPREGCOV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Politecnica de Madrid (Other)
Collaborators: Hospital Severo Ochoa (Other); Puerta de Hierro University Hospital (Other); Hospital Vall d'Hebron (Other); Hospital Universitario de Torrejón,Madrid (Other); Clínica Zuatzu de San Sebastián (Unknown)
Responsible Party: Principal Investigator, Rubén Barakat Carballo, Dr, Universidad Politecnica de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UPM-2020-32/33
Record Dates: First submitted 2020-09-19; First posted 2020-09-24 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Pregnancy Complications; Pregnancy, High Risk; Pregnancy Induced Hypertension; Newborn Morbidity; Fetal Growth Retardation; Fetus Disorder; Weight Gain, Maternal; Maternal-Fetal Relations
MeSH Terms: conditions — Pregnancy Complications; Hypertension, Pregnancy-Induced; Fetal Growth Retardation; Fetal Diseases; Gestational Weight Gain | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The design of the physical exercise program will be supported by the Canadian and Spanish Guidelines for exercise throughout pregnancy (11,13) and published by Barakat model (10).
  Frequency: The program will consist of three weekly sessions. The duration of every session will be 55-60 minutes. The intensity of the workload will be 55-60% of the maximum maternal Heart Rate, and controlled by Polar monitor (FT60). Likewise, once a week, the Borg Scale of Perceived Effort will be administered to participants, in order to have a more reliable assessment of the intensity of the activities, 12-14 (moderate; out of a 20 point scale) will be the level used.
  The minimum adherence required for the participants will be 80% of the total sessions (approximately 80 sessions).
  Interventions: Other: Exercise program; Other: Healthy lifestyle advise
- Control group (No Intervention): Women randomly assigned to the control group (CG) received general advice from their health care provider about the positive effects of physical activity. Participants in the CG had their usual visits with health care providers during pregnancy, which were equal to the exercise group. Women were not discouraged from exercising on their own. However, women in the CG were asked about their exercise once each trimester using a "Decision Algorithm" (by telephone).

INTERVENTIONS:
Other: Exercise program — All sessions will begin with a warm-up of 7-8 minutes composed of mild movements and joint mobility of upper and lower limbs exercises. Then a central part of 35-40 minutes, four types of activities will be included (aerobic work, muscle strengthening, coordination/balance tasks, pelvic floor exercises), finally a section of flexibility, relaxation and final talk (comments and sharing) will be performed (12-15 minutes).
  Arms: Exercise group
Other: Healthy lifestyle advise — This intervention consists of providing infographics and videos with advice on healthy habits throughout the pregnancy process. This type of content will be related to daily physical activity, food recommendations and fundamental exercises to perform during pregnancy.
  Arms: Exercise group

SUMMARY:
Historically and traditionally, the recommendations related to physical exercise during pregnancy have been based more on moral or cultural issues than on scientific evidence. During some phases of history, pregnancy has meant a period of seclusion for women (not only physical). One of the adverse consequences has been the common recommendation of rest as a general rule for pregnant women.

Scientific evidence from recent years has achieved a better understanding of the process of pregnancy and childbirth as well as maternal and fetal responses to exercise. Currently, both from a scientific and clinical/obstetric point of view, there is no doubt about the benefits of an active pregnancy for entire body of pregnant woman, and even her child. In fact, risks of a sedentary lifestyle are applicable to the pregnancy situation, even more with important associated complications during pregnancy and postpartum period.

Unfortunately, the impact of COVID-19 has caused an unprecedented global crisis, in this sense the necessary measures taken by the different administrations, especially in terms of confinement causes (from now on) a large number of complications affecting different populations. In summary a complex situation without established prevention strategies exists.

The pregnant population is, due to the nature of the gestation and delivery process, one of the population groups with the highest risk of adverse outcomes and associated complications and whose consequences include the mother, fetus, newborn and even children. According to an important body of scientific literature and based on an epigenetic effect, the intrauterine environment can be a determining factor for the future human being to evolve regardless of complications and pathologies (cardiovascular, metabolic, psychic, emotional). This is demonstrated by numerous recent scientific evidences that confirm the unfortunate association between an adverse intrauterine environment (due to various factors) and observable postnatal pathologies in infants.

In addition, current publications report the large number and variety of alterations that the COVID-19 situation causes in pregnant women and that includes the entire female organism. This complex situation does not only affect aspects of a physical or physiological nature, but also psychic and emotional factors. In summary, a new state of confinement or similar situations in the near future (impossibility of groupings, distance between people), avoid during the daily life of pregnant women one of the important and recent recommendations made by the international scientific community: a pregnancy physically active.

This is especially relevant, due to the dangerous association between complications of a psychological or emotional nature during pregnancy with pre, peri and postnatal disorders (low birth weights, perinatal complications, altered and prolonged deliveries, etc.), which affect not only to the mother and can determine the health of the future human being. According to the scientific literature and based on an epigenetic effect, the intrauterine environment can be a determining aspect in the health of the future human being and the prevention of complications and pathologies (cardiovascular, metabolic, psychic, emotional). This is demonstrated by numerous and recent scientific evidences that confirm the unfortunate association between an adverse intrauterine environment (due to various factors) and different pathologies during and after pregnancy.

It is evident the change that COVID-19 and its effects will generate in the lifestyle of the pregnant population and the increased probability of suffering associated pathologies in the next 24-36 months. No preventive actions have yet been planned in Spain and its public hospitals against the impact of COVID-19 on the quality of life of pregnant women. It is urgent to design and perform an adequate strategy of intervention for its possible prevention. From the scientific point of view, the recommendations are clear and concrete, an aerobic exercise program, designed and supervised by professionals from the Sciences of Physical Activity and Sports, is the best option for pregnant women.

In this sense, in the last 30 years, physical exercise has proven to have many benefits for pregnant women, without causing risks or adverse effects on maternal-fetal well-being. This is confirmed by an important body of scientific literature on gestational physical exercise and its effects on pregnancy outcomes.

DETAILED DESCRIPTION:
Hypothesis Aerobic, moderate, and supervised exercise during pregnancy can be an efficient element of prevention of alterations that the situation generated by COVID-19 causes to the healthy pregnant population and their children.

Objective Examine the influence of a supervised aerobic exercise program during pregnancy, by non-face-to-face and face-to-face ways, on the prevention of maternal, fetal, newborn and infant alterations during the pandemic state and in the near future.

Material and Methods

- Study design.

A randomized clinical trial (RCT) will be carried out, not masked with healthy pregnant women, giving rise to two study groups: exercise group (EG), pregnant women participating in a regular program of supervised physical exercise and control group ( CG), pregnant women who receive normal obstetric monitoring of their pregnancy, including recommendations regarding dietary-nutritional factors, as well as the benefits of an active pregnancy.

All selected pregnant women will sign an Informed Consent before participating in the study.

Women randomly assigned to the CG received general advice from their health care provider about the positive effects of physical activity. Participants in the CG had their usual visits with health care providers during pregnancy, which were equal to the exercise group. Women were not discouraged from exercising on their own. However, women in the CG were asked about their exercise once each trimester using a "Decision Algorithm" (by telephone).

Intervention

General characteristics of the physical exercise program:

* The minimum adherence required will be 80% of the total sessions.
* Onset: gestational week 9-11, immediately after the first prenatal ultrasound, in order to rule out Obstetric Contraindications for physical exercise.
* End: gestational week 38-39.
* Frequency: 3 weekly sessions, various possibilities will be offered at different times from which the pregnant woman can choose, in order to promote work and family conciliation.

Basic Considerations:

1. All the activity carried out will be aerobic.
2. Avoid working positions in which areas normally overloaded by pregnancy are further affected.
3. The work corresponding to flexibility will be carried out always bearing in mind that these are pregnant women, this forces us once again not to include forced operating positions in the exercises or to excessively maintain the stretching times in each area.
4. An adequate fluid intake will be maintained before and after the activity.
5. Also as a general rule and to eliminate potential risks, the following will be avoided:

   * Activities that include the Valsalva maneuver.
   * High ambient temperatures or very humid environments in order to avoid hyperthermia (body temperature higher than 38º C).
   * Sudden movements.
   * Positions of extreme muscular tension.

Structure:

All sessions will begin with a warm-up of 7-8 minutes composed of mild movements and joint mobility of upper and lower limbs exercises. Then a central part of 35-40 minutes, four types of activities will be included (aerobic work, muscle strengthening, coordination/balance tasks, pelvic floor exercises), finally a section of flexibility, relaxation and final talk (comments and sharing) will be performed (12-15 minutes).

Below we offer a greater detail of each part:

I. Warm-up-General activation. Displacements varied without impact activities (avoiding jumps, falls). Mild work of mobility of the main joints.

II. Aerobic section. Exercise to increase intensity up to moderate activities, play with sports equipment (balls, ropes, pikes) or choreographies of different musical styles.

III. Muscle strengthening, general toning exercises of the whole body: lower part (calf, quadriceps, hamstrings, adductors, abductors), upper part (abdominal, pectoral, shoulders, paravertebral musculature). Also exercises for the most weakened and needy muscle groups during pregnancy, the aim is to avoid muscular decompensation.

IV. Coordination and balance exercises: simple tasks of eye-hand and eye-foot coordination with sports equipment, as well as body axis balance exercises.

V. Strengthening the pelvic floor muscles, Kegel exercises will be applied and is basically composed of contractions (slow and fast) of the different structures of the pelvic floor musculature.

VI. Cool down section during 7-8 minutes, aiming to gradually lower the intensity of work with flexibility-stretching and relaxation exercises.

VII. Final Talk. This part is intended for pregnant women to express clearly and openly the sensations and perceptions experienced during the session. The reflection of each participant on the effect of physical practice is sought, not only in the physical or physiological aspect, but also in the psychic and emotional section. The exchange of impressions between the pregnant women, enhances the role of a correctly designed and conducted physical exercise program, as a social mobile of maintenance and improvement of the quality of life of the pregnant woman.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women fulfilling the following criteria: >18 years old, singleton pregnancies and planning management and delivery at the research hospitals and also do not participate in any other program of supervised physical exercise.

Exclusion Criteria:

* Women with absolute contraindications. Women with relative contraindications need permission from obstetric care provider prior to participation(1,2):

Absolute contraindications to exercise:

* Ruptured membranes.
* Premature labour.
* Unexplained persistent vaginal bleeding.
* Placenta praevia after 28 weeks' gestation.
* Pre-eclampsia.
* Incompetent cervix.
* Intrauterine growth restriction.
* High-order multiple pregnancy (eg, triplets).
* Uncontrolled type I diabetes.
* Uncontrolled hypertension.
* Uncontrolled thyroid disease.
* Other serious cardiovascular, respiratory or systemic disorder.

Relative contraindications to exercise:

* Recurrent pregnancy loss.
* Gestational hypertension.
* A history of spontaneous preterm birth.
* Mild/moderate cardiovascular or respiratory disease.
* Symptomatic anaemia.
* Malnutrition.
* Eating disorder.
* Twin pregnancy after the 28th week.
* Other significant medical conditions.

References:

1. Mottola, M. F., Davenport, M. H., Ruchat, S. M., Davies, G. A., Poitras, V. J., Gray, C. E., … Zehr, L. 2019 Canadian guideline for physical activity throughout pregnancy. British Journal of Sports Medicine, 2018; 52(21), 1339-1346. https://doi.org/10.1136/bjsports-2018-100056.
2. Barakat R, Díaz-Blanco A, Franco E, Rollán-Malmierca A, Brik M, Vargas M, et al. Guías clínicas para el ejercicio físico durante el embarazo/Clinical guidelines for physical exercise during pregnancy. Prog Obstet Ginecol 2019;62(5):464-471. DOI: 10.20960/j.pog.00231.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal weight gain | 9 months
  analyze the increase during pregnancy
blood pressure | 9 months
  analyze how it varies during pregnancy
OGTT-O'Sullivan test | 1 month
  analyze the value and its interrelationship with physical exercise patterns
Urinary Incontinence Questionnaire (ICIQ-SF) | 9 months
  analyze with a questionnaire the value and its interrelationship with physical exercise patterns (different measures in the questionnaire)
State-Trait Anxiety Inventory (STAI) | 9 months
  analyze with a questionnaire the value and its interrelationship with physical exercise patterns (Likert scale 0-3)
depression scale (CES-D) | 9 months
  analyze with a questionnaire the variability during pregnancy (Likert scale 0-3)
Behavior of Fetal Heart Rate | 3 months
  analyze variability during pregnancy
gestational age | 9 months
  analyze the value and its interrelationship with physical exercise patterns
type of delivery (Vaginal, instrumental or cesarean) | 1 month
  analyze whether women have had a vaginal, instrumental or cesarean delivery and its interrelationship with physical exercise patterns
duration of labor | 1 month
  analyze the value and its interrelationship with physical exercise patterns
birthweight | 1 month
  analyze the value and its interrelationship with physical exercise patterns
child's weight | 24 months
  analyze the value and its interrelationship with physical exercise patterns during pregnancy
child's height | 24 months
  analyze the value and its interrelationship with physical exercise patterns during pregnancy
mental assessment of the child (depression questionnaire adapted to childhood) | 24 months
  analyze the value and its interrelationship with physical exercise patterns during pregnancy (Likert scale 0-3)
psychomotor behavior of the child | 24 months
  analyze some variables (sitting, crawling, standing, walking, holding objects...) and its relationship with maternal exercise

SECONDARY OUTCOMES:
Maternal pains during pregnancy (headache, back pain, pelvic pain, paravertebral, scapular, etc.) | 9 months
  analyze the value and its interrelationship with physical exercise patterns
fetal growth and development | 9 months
  analyze the value and its interrelationship with physical exercise patterns
Delivery tears | 1 month
  analyze the value and its interrelationship with physical exercise patterns
performing episiotomy during childbirth | 1 month
  analyze the appearance (descriptive: yes/no) and its interrelationship with physical exercise patterns
Apgar Score | 1 month
  analyze the value and its interrelationship with physical exercise patterns
length | 1 month
  analyze the value and its interrelationship with physical exercise patterns
cranial perimeter | 1 month
  analyze the value and its interrelationship with physical exercise patterns
Landau reflexes test | 1 month
  analyze the value and its interrelationship with physical exercise patterns
neonatal intensive care unit (NICU) | 1 month
  analyze the number of admissions and its interrelationship with physical exercise patterns
Postpartum recovery of pre-pregnancy weight | 12 months
  analyze how it varies during postpartum period
Edinburgh Postpartum Depression Scale (EPDS) | 12 months
  analyze with a questionnaire how it varies during postpartum period (Likert scale 0-3)
umbilical cord Ph | 1 month
  analyze the value and its interrelationship with physical exercise patterns
Fetal development | 9 months, once a trimester
  analyze variables (estimated fetal weight, FCF, DBT, CRL, SNT, uterine arteries...) by ultrasound
Carotid intima-media thickness (CIMT) | 9 months
  Measurement of carotid intima-media thickness (CIMT) with B-mode ultrasound is a noninvasive, sensitive, and reproducible technique for identifying and quantifying subclinical vascular disease and for evaluating CVD risk.
Maternal sleep habits | 9 months
  analyze with Pittsburgh´s sleep quality index
maternal body self-perception | 9 months
  analyze using Ben-Tobim Walker Body Attitude Questionnaire
Newborn sleep habits | 24 months
  analyze using Brief Infant Sleep Questionnaire
Placental angiogenic factors | measured at 24-25 weeks and at 34-35 weeks
  placental growth factor (PIGF)
Placental angiogenic factors | measured at 24-25 weeks and at 34-35 weeks
  soluble fms-like tyrosinekinase-1(sFlt1)
Lipidic profile | measured at 24-25 weeks and at 34-35 weeks
  Total Cholesterol, LDL-Cholesterol, HDL- Cholesterol, Tryglicerids

OTHER OUTCOMES:
Perception of health status - SF36 health scale | 24 months
  analyze the value and its interrelationship with physical exercise patterns (Likert scale)
Recovery of pelvic floor muscles ultrasound | 6 months
  analyze the diameter and thickness of muscles in the perineal area and its interrelationship with physical exercise patterns
Maternal habits of physical activity - Pregnancy Physical Activity Questionnaire (PPAQ) | 12 months
  analyze with a questionnaire how it varies during and after pregnancy
Pregestational maternal patterns | 9 months
  analyze sociodemographic and behavioural habits like (smoking, alcoholism, pervious illness, COVID-19, parity, occupation, previous miscarriage...)
Edimburgh postpartum depression scale | 6 months
  analyze with a questionnaire the variability in the postpartum
Covid-19 disease | 9 months
  analyze the covid-19 condition durign pregnancy and its interrelationship with other variables

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Barakat, Dr, Study Director — Universidad Politécnica de Madrid (UPM)
Locations (2):
- Spain (2):
  - Facultad de Ciencias de la Actividad Física y el Deporte (INEF), Madrid
  - Facultad de Ciencias de la Actividad Física y el Deporte - INEF, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barakat R, Pelaez M, Cordero Y, Perales M, Lopez C, Coteron J, Mottola MF. Exercise during pregnancy protects against hypertension and macrosomia: randomized clinical trial. Am J Obstet Gynecol. 2016 May;214(5):649.e1-8. doi: 10.1016/j.ajog.2015.11.039. Epub 2015 Dec 15. PMID 26704894
- [Background] Barakat R, Franco E, Perales M, Lopez C, Mottola MF. Exercise during pregnancy is associated with a shorter duration of labor. A randomized clinical trial. Eur J Obstet Gynecol Reprod Biol. 2018 May;224:33-40. doi: 10.1016/j.ejogrb.2018.03.009. Epub 2018 Mar 6. PMID 29529475
- [Background] Barakat R, Refoyo I, Coteron J, Franco E. Exercise during pregnancy has a preventative effect on excessive maternal weight gain and gestational diabetes. A randomized controlled trial. Braz J Phys Ther. 2019 Mar-Apr;23(2):148-155. doi: 10.1016/j.bjpt.2018.11.005. Epub 2018 Nov 17. PMID 30470666
- [Background] Vargas-Terrones M, Nagpal TS, Barakat R. Impact of exercise during pregnancy on gestational weight gain and birth weight: an overview. Braz J Phys Ther. 2019 Mar-Apr;23(2):164-169. doi: 10.1016/j.bjpt.2018.11.012. Epub 2018 Nov 22. PMID 30527949
- [Background] Fernandez-Buhigas I, Brik M, Martin-Arias A, Vargas-Terrones M, Varillas D, Barakat R, Santacruz B. Maternal physiological changes at rest induced by exercise during pregnancy: A randomized controlled trial. Physiol Behav. 2020 Jun 1;220:112863. doi: 10.1016/j.physbeh.2020.112863. Epub 2020 Mar 8. PMID 32160968
- [Background] Mourtakos SP, Tambalis KD, Panagiotakos DB, Antonogeorgos G, Arnaoutis G, Karteroliotis K, Sidossis LS. Maternal lifestyle characteristics during pregnancy, and the risk of obesity in the offspring: a study of 5,125 children. BMC Pregnancy Childbirth. 2015 Mar 21;15:66. doi: 10.1186/s12884-015-0498-z. PMID 25885759
- [Background] Contreras ZA, Ritz B, Virk J, Cockburn M, Heck JE. Maternal pre-pregnancy and gestational diabetes, obesity, gestational weight gain, and risk of cancer in young children: a population-based study in California. Cancer Causes Control. 2016 Oct;27(10):1273-85. doi: 10.1007/s10552-016-0807-5. Epub 2016 Sep 9. PMID 27613707
- [Background] Badon SE, Littman AJ, Chan KCG, Tadesse MG, Stapleton PL, Bammler TK, Sorensen TK, Williams MA, Enquobahrie DA. Physical activity and epigenetic biomarkers in maternal blood during pregnancy. Epigenomics. 2018 Nov;10(11):1383-1395. doi: 10.2217/epi-2017-0169. Epub 2018 Oct 16. PMID 30324807
- [Background] Shrestha D, Workalemahu T, Tekola-Ayele F. Maternal dyslipidemia during early pregnancy and epigenetic ageing of the placenta. Epigenetics. 2019 Oct;14(10):1030-1039. doi: 10.1080/15592294.2019.1629234. Epub 2019 Jun 14. PMID 31179827
- [Background] Physical Activity and Exercise During Pregnancy and the Postpartum Period: ACOG Committee Opinion, Number 804. Obstet Gynecol. 2020 Apr;135(4):e178-e188. doi: 10.1097/AOG.0000000000003772. PMID 32217980
- [Background] Mottola MF, Davenport MH, Ruchat SM, Davies GA, Poitras VJ, Gray CE, Jaramillo Garcia A, Barrowman N, Adamo KB, Duggan M, Barakat R, Chilibeck P, Fleming K, Forte M, Korolnek J, Nagpal T, Slater LG, Stirling D, Zehr L. 2019 Canadian guideline for physical activity throughout pregnancy. Br J Sports Med. 2018 Nov;52(21):1339-1346. doi: 10.1136/bjsports-2018-100056. PMID 30337460
- [Background] Barakat R. An exercise program throughout pregnancy: Barakat model. Birth Defects Res. 2021 Feb 1;113(3):218-226. doi: 10.1002/bdr2.1747. Epub 2020 Jul 2. PMID 32613735
- [Background] Yang Z, Wang M, Zhu Z, Liu Y. Coronavirus disease 2019 (COVID-19) and pregnancy: a systematic review. J Matern Fetal Neonatal Med. 2022 Apr;35(8):1619-1622. doi: 10.1080/14767058.2020.1759541. Epub 2020 Apr 30. PMID 32354293
- [Background] Della Gatta AN, Rizzo R, Pilu G, Simonazzi G. Coronavirus disease 2019 during pregnancy: a systematic review of reported cases. Am J Obstet Gynecol. 2020 Jul;223(1):36-41. doi: 10.1016/j.ajog.2020.04.013. Epub 2020 Apr 18. PMID 32311350
- [Background] Novakovic B, Saffery R. The ever growing complexity of placental epigenetics - role in adverse pregnancy outcomes and fetal programming. Placenta. 2012 Dec;33(12):959-70. doi: 10.1016/j.placenta.2012.10.003. Epub 2012 Oct 24. PMID 23102655
- [Background] Khan S, Jun L, Nawsherwan, Siddique R, Li Y, Han G, Xue M, Nabi G, Liu J. Association of COVID-19 with pregnancy outcomes in health-care workers and general women. Clin Microbiol Infect. 2020 Jun;26(6):788-790. doi: 10.1016/j.cmi.2020.03.034. Epub 2020 Apr 8. No abstract available. PMID 32278081
- [Background] Perales M, Valenzuela PL, Barakat R, Cordero Y, Pelaez M, Lopez C, Ruilope LM, Santos-Lozano A, Lucia A. Gestational Exercise and Maternal and Child Health: Effects until Delivery and at Post-Natal Follow-up. J Clin Med. 2020 Jan 31;9(2):379. doi: 10.3390/jcm9020379. PMID 32023833
- [Background] Pelaez M, Gonzalez-Cerron S, Montejo R, Barakat R. Protective Effect of Exercise in Pregnant Women Including Those Who Exceed Weight Gain Recommendations: A Randomized Controlled Trial. Mayo Clin Proc. 2019 Oct;94(10):1951-1959. doi: 10.1016/j.mayocp.2019.01.050. PMID 31585579
- [Background] Perales M, Refoyo I, Coteron J, Bacchi M, Barakat R. Exercise during pregnancy attenuates prenatal depression: a randomized controlled trial. Eval Health Prof. 2015 Mar;38(1):59-72. doi: 10.1177/0163278714533566. Epub 2014 May 28. PMID 24872442
- [Background] Barakat R, Perales M, Garatachea N, Ruiz JR, Lucia A. Exercise during pregnancy. A narrative review asking: what do we know? Br J Sports Med. 2015 Nov;49(21):1377-81. doi: 10.1136/bjsports-2015-094756. Epub 2015 Jul 1. PMID 26135742
- [Derived] Martin-Arias A, Fernandez-Buhigas I, Aramburu-Anglada C, Pino AA, Saez RB, Rolle V, Sanchez-Polan M, Silva-Jose C, Gil MM, Santacruz B. The Effect of a Supervised Exercise Program Throughout Pregnancy on Longitudinal Lipid Profile Changes: A Randomized Clinical Trial. Matern Fetal Med. 2026 Jan;8(1):40-47. doi: 10.1097/FM9.0000000000000318. Epub 2025 Sep 26. PMID 41624594
- [Derived] Zhang D, Sanchez-Polan M, Silva-Jose C, Diaz-Blanco A, Brik M, Arias AM, Hernando P, Barakat R. Prenatal Exercise Decreases Urinary Incontinence in Late Pregnancy and 3 Months Postpartum: A Randomized Controlled Trial. Med Sci Sports Exerc. 2025 Mar 1;57(3):555-562. doi: 10.1249/MSS.0000000000003597. Epub 2024 Nov 18. PMID 39809234
- [Derived] Uria-Minguito A, Silva-Jose C, Sanchez-Polan M, Diaz-Blanco A, Garcia-Benasach F, Carrero Martinez V, Alzola I, Barakat R. The Effect of Online Supervised Exercise throughout Pregnancy on the Prevention of Gestational Diabetes in Healthy Pregnant Women during COVID-19 Pandemic: A Randomized Clinical Trial. Int J Environ Res Public Health. 2022 Oct 28;19(21):14104. doi: 10.3390/ijerph192114104. PMID 36360995
- See also: Reference of the Spanish clinical guidelines of physical exercise for pregnancy — https://dialnet.unirioja.es/servlet/articulo?codigo=7357988